CLINICAL TRIAL: NCT00998881
Title: A Phase III, Double-blind, Placebo Controlled, Monotherapy Study of MP-513 in Japanese Patients With Type 2 Diabetes Mellitus - Confirmative Study
Brief Title: Monotherapy Study of MP-513 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3000-A5
Record Dates: First submitted 2009-10-15; First posted 2009-10-21 (Estimated); Results first posted 2014-02-21 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teneligliptin 20 mg (Experimental): Teneligliptin 20 mg, orally, once daily
  Interventions: Drug: Teneligliptin 20 mg
- Placebo (Placebo Comparator): Teneligliptin placebo-matching tablets, orally, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Teneligliptin 20 mg
  Other Names: MP-513
  Arms: Teneligliptin 20 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of MP-513 (Teneligliptin) in patients with type 2 Diabetes for 12 weeks administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 20 - 75 years old
* Patients who are under dietary management and taking therapeutic exercise for diabetes over 12 weeks before administration of investigational drug
* Patients whose HbA1c is between 6.5% - 10.0%
* Patients who were not administered diabetes therapeutic drugs within 12 weeks before administration of investigational drug.

Exclusion Criteria:

* Patients with type 1 diabetes, diabetes mellitus caused by pancreas impairment, or secondary diabetes (Cushing disease, acromegaly, etc)
* Patients with Class III/IV heart failure symptoms according to New York Heart Association (NYHA) functional classification
* Patients with serious diabetic complications.
* Patients who are habitual excessive alcohol consumption.
* Patients with severe hepatic disorder or severe renal disorder.
* Patients who are pregnant, lactating, and probably pregnant patients, and patients who can not agree to contraception

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Kadowaki, Professor, Study Director — Tokyo University; Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation
Locations (1):
- Sapporo, Hokkaido, Japan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Teneligliptin 20 mg
Started | 104 | 99
Completed | 96 | 97
Not Completed | 8 | 2
Not completed — Adverse Event | 2 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Personal matter | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Teneligliptin 20 mg | Total
Number analyzed (Participants) | 104 | 99 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (10.1) | 58.5 (10.0) | 58.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 31 | 65
  Male | 70 | 68 | 138

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 12
Description: The change from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Week 12. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline HbA1c as a covariate.
Time Frame: 12 weeks
Population: The full analysis set, consisting of all type 2 diabetic patients, who received at least one dose of study drug and who had at least one efficacy data after randomization. Analysis based on last observation carried forward, where the last postbaseline double-blind observed value was carried forward and used for Week 12 where data was missing.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Teneligliptin 20 mg
Number analyzed (Participants) | 104 | 99
Percent | 0.17 (0.05) | -0.62 (0.05)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 12
Description: The change from Baseline in Fasting Plasma Glucose collected at Week 12. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline Fasting Plasma Glucose as a covariate.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg / dL
Arm/Group | Placebo | Teneligliptin 20 mg
Number analyzed (Participants) | 104 | 99
mg / dL | -0.2 (1.8) | -19.2 (1.8)

3. Secondary Outcome: Change From Baseline in the Areas Under the Curve From 0 to 2 h (AUC0-2h) for Postprandial Plasma Glucose at Week 12
Description: The change from Baseline in AUC0-2h for Postprandial Plasma Glucose collected at Week 12. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline AUC0-2h for Postprandial Plasma Glucose as a covariate.
Time Frame: 12 weeks
Population: The full analysis set, consisting of all type 2 diabetic patients, who received at least one dose of study drug and who had at least one efficacy data after randomization.
Measure: Least Squares Mean (Standard Error); unit: mg*h / dL
Arm/Group | Placebo | Teneligliptin 20 mg
Number analyzed (Participants) | 96 | 97
mg*h / dL | 0.224 (4.849) | -73.124 (4.824)

4. Secondary Outcome: Change From Baseline in 2-hour Postprandial Plasma Glucose at Week 12
Description: The change from Baseline in 2-hour Postprandial Plasma Glucose collected at Week 12. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline 2-hour Postprandial Plasma Glucose as a covariate.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mg / dL
Arm/Group | Placebo | Teneligliptin 20 mg
Number analyzed (Participants) | 96 | 97
mg / dL | -3.2 (3.6) | -47.9 (3.5)

ADVERSE EVENTS:
Arm/Group | Placebo | Teneligliptin 20 mg
Serious Adverse Events (participants affected / at risk) | 4/104 | 0/99
Other Adverse Events (participants affected / at risk) | 63/104 | 62/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=104) | Teneligliptin 20 mg (N=99)
Vestibular neuronitis (Infections and infestations) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=104) | Teneligliptin 20 mg (N=99)
Acute sinusitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 4 | 3
Cystitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 3 | 2
Hordeolum (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 7 | 12
Pharyngitis (Infections and infestations) | 1 | 1
Tinea pedis (Infections and infestations) | 3 | 0
Helicobacter infection (Infections and infestations) | 0 | 1
Alveolar osteitis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 2
Anxiety disorder (Psychiatric disorders) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Blepharospasm (Eye disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Colonic polyp (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 2 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Periodontitis (Gastrointestinal disorders) | 4 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 2
Gastric xanthoma (Gastrointestinal disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Micturition disorder (Renal and urinary disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Feeling abnormal (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Vessel puncture site haematoma (General disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood creatine phosphokinase increased (Investigations) | 4 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 4 | 0
Blood urea increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 1 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Glucose urine present (Investigations) | 7 | 4
Blood urine present (Investigations) | 3 | 2
White blood cell count increased (Investigations) | 0 | 2
Protein urine present (Investigations) | 3 | 2
Urine ketone body present (Investigations) | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Mouth injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other